CLINICAL TRIAL: NCT03892343
Title: A Prospective Study of the Effects of Renal Transplantation on Uraemic Cardiomyopathy Using Magnetic Resonance Imaging.
Brief Title: Effects of Renal Transplantation on Uraemic Cardiomyopathy
Acronym: RETRACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Charles Ferro, Dr, Professor Charles Ferro, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: RRK6458
Record Dates: First submitted 2019-02-27; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cardiomyopathies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Markers of CKD-MBD: - calcium, phosphate, alkaline phosphatase and PTH will be analyzed in serum by mass spectroscopy and FGF-23 will be analyzed by ELISA at 0 and 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transplant recipients: Patients undergoing live donor kidney transplant.
  Interventions: Diagnostic Test: Cardiac MRI
- Non-transplanted: Patients on the deceased donor waiting list without prospect of a live donor transplant.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac Magnetic Resonance Imaging (Siemens Skyra 3T): will be performed using protocols and techniques already in use in our group. All CMR scan derived parameters will be analysed with the investigator blinded to treatment allocation as in previous studies.

SUMMARY:
Chronic kidney disease (CKD) is associated with a high risk of death and morbidity due to cardiovascular disease. Much of this is caused by left ventricular disease characterised by abnormal muscle thickness and scaring. This process appears to start early in the course of CKD and causes heart failure and dangerous abnormal heart rhythms. Previous work suggests that the process may be reversible by kidney transplantation but almost all of the studies are small, retrospective and lack scientific rigour. Furthermore, they almost all use echocardiography, which is inaccurate in patients with CKD. The investigators plan to perform the first large, prospective, controlled, blind-analysed study using cardiac magnetic resonance imaging to determine whether CKD associated cardiomyopathy is reversed by kidney transplantation and if so, whether factors such as blood pressure and mediators of metabolic bone disease/fibrosis are important in effecting this change. Greater understanding of the mechanisms responsible for CKD associated cardiomyopathy could lead to future strategies and treatments to improve the high cardiovascular mortality associated with this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients registered on the kidney transplant waiting list at the University Hospital Birmingham NHS Foundation Trust.
2. Ages over 18 years

Exclusion Criteria

1. Non-standard anti-rejection treatment, post transplant.
2. Previous history of being unable to tolerate MRI scanner.
3. Contraindication to MRI - eg metal fragments in ey

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise of patients with end-stage renal failure currently awaiting either live or deceased donor transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Mass | One year.
  Calculated by Cardiac MRI

SECONDARY OUTCOMES:
Native Myocardial T1 Times. | One year.
  Measured using T1 mapping techniques (MOLLI)
Blood Pressure | One year.
  24hr Ambulatory Blood pressure monitoring
Pulse Wave Analysis. | One Year
  To calculate augmentation index as a marker of arterial stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ferro, MD, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- Queen Elizabeth Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No